CLINICAL TRIAL: NCT05707000
Title: Comparison of Concentric Quadriceps Strengthening and Facilitatory Kinesiotaping on Gait Parameters in Knee Osteoarthritis
Brief Title: Comparison of Quadriceps Strengthening and Kinesiotaping on Gait in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RiphahIU farhana Nasir
Record Dates: First submitted 2023-01-22; First posted 2023-01-31 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis; Quadriceps; Kinesiotaping
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A, Concentric Muscle Training (Experimental): leg press, knee flexion, knee extension, Quad drills with 1 RM
  Interventions: Other: group A concentric muscle training
- group B, Quadriceps Facilitatory Kinesiotaping (Experimental): kinesiotaping on the quadriceps muscle in the faciliatory mode
  Interventions: Other: Group B fascilitatory kinesiotaping

INTERVENTIONS:
Other: group A concentric muscle training — One set of each of the following exercises will completed during each session:
  * leg press,
  * knee flexion,
  * knee extension,
  * Quad drills For each set, 12 repetitions will be performed at a resistance load of 60% of the one-repetition maximum (1RM) for that exercise. The exercises will be performed 2 times a week for 6 weeks.
  Arms: group A, Concentric Muscle Training
Other: Group B fascilitatory kinesiotaping — Kinesiotaping is applied on the anterior thigh (quadriceps) region starting at 1/5 of the distance between anterosuperior iliac spine (ASIS) and tibia tuberosity. The tape is applied with 20% tension of the tape. The tape was tensioned from proximal region of mid quadriceps down to tibia tuberosity and, once it reached the knee, the tape was divided in the middle allowing it to circle the joint
  Arms: group B, Quadriceps Facilitatory Kinesiotaping

SUMMARY:
The aim of this research is to determine the Effects of facilitatory Kinesio-taping and concentric quadriceps strengthening on gait parameters in knee osteoarthritis. Randomized clinical trials will be done at Physio Experts Clinic, Islamabad. The sample size is 38. The subjects were divided in two groups, with 19 subjects in Group A and 19 in Group B. Study duration was of 6 months. Sampling technique applied was Non probability Convenience Sampling technique. Both males and females of aged 50-60 years with Knee OA grade 2 or 3 were included. Tools used in the study are Numeric Pain Rating Score (NPRS), dynamometer, WOMAC questionnaire and Mobile app for measuring Temporospatial gait parameters.

DETAILED DESCRIPTION:
Osteoarthritis is one of the most common musculoskeletal disorders in adults. It is a degenerative joint disease affecting 15%-40% of people more than 40 years of age. The term osteoarthritis was authored in 1886 by the English doctor, John Kent Spender. Clinical assessment to recognize OA from RA and other comparable conditions turned out to be broadly acknowledged by the main decade of the twentieth century enormous because of the endeavors set forward by Archibald E.

Osteoarthritis is a degenerative joint condition that causes other joint tissues to lose gross cartilage and to experience morphological damage. Pathological changes seen in knee osteoarthritis joints include progressive loss and destruction of articular cartilage, thickening of the subchondral bone, formation of osteophytes, variable degrees of inflammation of the synovium, degeneration of ligaments and menisci of the knee and hypertrophy of the joint capsule. Biomechanical factor that is assumed to contribute to the etiology of OA is laxity of knee joint, which is described as the rotation or displacement of femur from tibia. One research found that Varus-valgus laxity in patients with unaltered knees and unilateral OA is wider than in stable healthy participants, indicating knee joint laxity may be disease predisposing. the progress of the lateral and medial knee OA, as defined by narrowing of joint space and a degradation of physical activity, was found to have been linked with lower limb valgus-Varus alignment.

The main focus in OA management is on promoting self-management, reducing pain, optimize function, and modifying the disease process and its effects. The primary treatment for OA knee conservatively is physiotherapy which includes strength training, modalities, knee bracing, resistance training and Kinesiotaping. Resistance exercise can reduce knee pain severity and leg strength in participants with symptomatic knee OA. Exercise interventions using free weights or machines have generally focused on movements with concentric muscle contractions. Previous interventions were developed based on loads lifted during the concentric phase.

Kinesiotape (KT), is an elastic woven-cotton strip with a heat- sensitive acrylic adhesive structure.

ELIGIBILITY:
Inclusion Criteria:

* Adults of age 50- 60 years
* Presence of OA of the knee (using American College of Rheumatology criteria) for ≥6 months
* Knee pain due to tibiofemoral knee OA not from Patellofemoral OA
* Bilateral standing anterior-posterior radiograph demonstrating Kellgren and Lawrence OA grade 2 or 3

Exclusion Criteria:

* Knee surgery within last 12 months
* Lumber radiculopathy
* Vascular claudication
* Anterior knee pain due to diagnosed Patellofemoral syndrome/ chondromalacia
* Administered corticosteroid or hyaluronic injections within 3 months
* Any other MSK limitations
* Any cardiovascular problems

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Temporo-spatial Gait Parameters: | 6 week
  Measurement of temporospatial gait parameters (gait velocity, cadence, step length, step width and single support time) and their assessment, and calculating normalized values using the mobile app

SECONDARY OUTCOMES:
Numeric Pain Rating Score (NPRS): | 6 week
  Pain due to Knee OA was assessed using a numerical pain rating scale (NPRS), and scoring range 0, no pain, to 10, maximum pain.
Functional Status (WOMAC Questionnaire): | 6 week
  Functional Status is measured using WOMAC questionnaire. The WOMAC is a self-reported, lower extremity specific questionnaire and contains 24 questions: 17 on physical function, 5 on pain, and 2 on stiffness.
Strength | 6 week
  Strength is calculated using hand held dynamometer that offers a reliable and valid method to quantify quadriceps strength in a clinical environment

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Razzaq, MSPT-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Physio Experts Clinic, Islamabad, Capital, Pakistan

IPD SHARING:
Plan to Share IPD: No